CLINICAL TRIAL: NCT05325112
Title: ADVANCE-ED: Assessing Diagnostic Value of Non-invasive FFR-CT in Coronary Care in the Emergency Department
Brief Title: Assessing Diagnostic Value of Non-invasive FFR-CT (Fractional Flow Reserve - Computed Tomography) in Coronary Care in the Emergency Department
Acronym: ADVANCE-ED
Status: Terminated | Type: Observational
Why Stopped: Sponsor decision to terminate the study
Sponsor: HeartFlow, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CP- 909-001
Record Dates: First submitted 2022-04-05; First posted 2022-04-13 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- FFR-CT Group: Sites who have CCTA and FFR-CT analysis incorporated into their standard evaluation of chest pain in the ED/observation unit.
  Interventions: Diagnostic Test: FFRCT
- Control Group: Sites who have CCTA but not FFR-CT incorporated into the ED/observation unit.

INTERVENTIONS:
Diagnostic Test: FFRCT — FFRCT is a diagnostic test following a CCTA to help diagnose and treat coronary artery disease.
  Groups: FFR-CT Group

SUMMARY:
This is a prospective multi-center study. All clinically stable, symptomatic patients who present to the emergency department (ED) or observation unit with suspected coronary artery disease (CAD) and who have at least one ≥40% lesion and no lesion >90% confirmed by CCTA (Coronary Computed Tomography Angiogram) are eligible for enrollment once their CCTA has been completed and their FFR-CT (if applicable) has been ordered. All enrolling sites will have CCTA incorporated into their standard evaluation of chest pain in the ED/observation unit. Non-control sites will have CCTA and FFR-CT analysis incorporated into their standard evaluation of chest pain in the ED/observation unit.

DETAILED DESCRIPTION:
This is a prospective multi-center study. All clinically stable, symptomatic patients who present to the ED or observation unit with suspected CAD and who have at least one ≥40% lesion and no lesions <90% lesion in a major vessel, confirmed by CCTA, are eligible for enrollment once their CCTA has been completed and FFR-CT (if applicable) has been ordered. All enrolling sites will have CCTA incorporated into their standard evaluation of chest pain in the ED/observation unit. Non-control sites will have CCTA and FFR-CT analysis incorporated into their standard evaluation of chest pain in the ED/observation unit.

All participating sites will provide demographics, medical history, CCTA images, FFR-CT (for non-control sites), the decision plan post CCTA and pre FFR-CT (for non-control sites), length of stay for patients in the ED/observation unit/hospital, billing reports (UB-04 preferred), 30-day clinical outcomes, and any other hospital or office visits, imaging, and/or procedural data completed prior to the follow-up 30-day visit. Sites which do not have FFR-CT incorporated into the ED/observation unit will be control sites.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Clinically stable, symptomatic patients who present to ED/observation unit with suspected CAD
3. CCTA shows at least one ≥40% lesion and no lesions >90% in at least one major epicardial vessel
4. FFR-CT processed successfully (if applicable)
5. EKG with no acute ischemic changes
6. Willing to comply with all aspects of the protocol, including adherence to follow up visit
7. Agrees to be included in the study
8. Able to provide written informed consent

Exclusion Criteria:

1. CCTA showing no ≥40% lesion in a major epicardial vessel
2. CCTA showing a lesion >90% in a major epicardial vessel
3. CCTA showing other incidental, non-cardiac findings requiring admission, e.g., pneumonia, pulmonary embolism, or aortic dissection
4. Uninterpretable CCTA which is not of diagnostic quality
5. Coronary artery bypass graft surgery (CABG) or percutaneous coronary intervention (PCI) prior to CCTA acquisition
6. Left main lesion >50%
7. Confirmed acute coronary syndrome (acute myocardial infarction or unstable angina)
8. Known complex congenital heart disease or any history of coronary artery disease
9. Patients with tachycardia or significant arrhythmia which cannot be adequately controlled with medications to allow CTA
10. Any active, serious, life-threatening disease with a life expectancy of less than 2 months
11. Inability to comply with follow-up requirements
12. Currently enrolled in another study utilizing FFR-CT or in an investigational trial that involves a non-approved cardiac drug or device
13. Persons under the protection of justice, guardianship, or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinically stable, symptomatic patients who present to the ED with suspected coronary artery disease and no history of coronary artery disease, and who while in the ED have a CCTA performed which shows at least one ≥40% lesion and no lesions >90% in a major epicardial vessel, and a successfully processed FFR-CT (if applicable).
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2022-07-15 (Actual); Primary Completion 2022-11-14 (Actual); Study Completion 2022-11-14 (Actual)

PRIMARY OUTCOMES:
Reclassification rate between the coronary management plan based on the review of the CCTA alone compared to the coronary management plan based on the review of the CCTA and the FFR-CT analysis. | 30 days

SECONDARY OUTCOMES:
Cost Utility Analysis | 30 days
  Cost measurements to include length of stay in the emergency department and in the hospital overall, secondary coronary artery disease testing, and invasive procedures done.
Rate of Major Adverse Coronary Events (MACE) | 30 days
Time to primary diagnosis | Within 30 days
  Time between when the patient first arrives to the emergency department to when the treating physician documents the primary diagnosis.
Time to discharge | Within 30 days
  Time between when the patient first arrives to the emergency department to the time the patient was discharged from the emergency department or the hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Sadeer Al-Kindi, MD, Principal Investigator — University Hospitals Cleveland; Sneha Chinai, MD, Principal Investigator — UMass Memorial Health
Locations (2):
- United States (2):
  - UMass Memorial Hospital, Worcester, Massachusetts
  - University Hospital Clevelan, Cleveland, Ohio